CLINICAL TRIAL: NCT06131502
Title: ExAblate MR-guided Focused Ultrasound Bilateral Anterior Capsulotomy for Treatment of Obsessive-Compulsive Disorder
Brief Title: Sonication-based OCD Neurosurgical Intervention Via Capsulotomy
Acronym: SONIC
Status: Suspended | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: The IRB for this project lapsed, the IDE transfer to Dr. Joseph Taylor is underway, and there may be a possible change in funding source. Pending IRB re-submission in 2026.
Sponsor: Brigham and Women's Hospital (Other)
Collaborators: Stanford University (Other)
Responsible Party: Principal Investigator, Joseph J. Taylor, MD, PhD, Principal Investigator, Brigham and Women's Hospital
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 2023P002879
Record Dates: First submitted 2023-11-09; First posted 2023-11-14 (Actual); Last update posted 2025-10-29 (Actual); Status verified 2025-10

CONDITIONS: Obsessive-Compulsive Disorder
Keywords: OCD; neuroimaging; neurosurgery; MR-guided focused ultrasound (MRgFUS); Capsulotomy
MeSH Terms: conditions — Obsessive-Compulsive Disorder

STUDY DESIGN:
Intervention Model Description: In the first stage of the study, participants with severe, treatment resistant OCD (n=10) will be recruited in two centers (Harvard and Stanford) and treated with best medical care (BMT) for 6 months. Thereafter, they will receive the ExAblate MRgFUS procedure and then another BMT for 12 months. In the second stage of the study, participants with moderate to severe OCD (n=56) will be recruited in a multi-center study and treated with BMT plus real or sham MRgFUS for 12 months. Thereafter, those who received sham MRgFUS and did not improve will receive real MRgFUS and then treated with BMT for another 12 months.
Who Masked: Participant, Outcomes Assessor
Masking Description: In the first stage, patients will not be randomized and neither patients nor evaluators will be blinded as to treatment status. A period of 6 months of best medical treatment (BMT) prior to the capsulotomy treatment will ensure that the patients are clinically stable and compliant with the study set-up.
  If no safety stop rules occur at the end of the first stage, we will submit an IDE supplement to the FDA providing evidence of safety and requesting continuation. The second stage would then proceed pending the receipt and review/approval of that supplement. The second stage is focused on efficacy. In stage II, patients will be randomized, and both patient and evaluators will be blinded as to treatment status. The patients will be treated by BMT plus MRgFUS or BMT plus sham for 12 months. Parallel BMT along with the sham and MRgFUS periods would decrease protocol violations or drop-outs.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Real FUS (Active Comparator): The treatment volume and plan will be defined by the neurosurgeon. The ExAblate MRgFUS system will automatically compute the number of sonications, and the (per sonication spot) phase and amplitude corrections necessary for the system to produce a focal spot at each of the desired locations. The target selected for this study is the anterior limb of the internal capsule (ALIC). The target will be approximately 7-10mm rostral to the anterior edge of the anterior commissure, in the ventral part of the ALIC. A central point in the targeted area will be targeted with a low dose, sub-lethal energy level sonication to confirm the targeting accuracy on the MR images. Focal point position and/or transducer location will be adjusted as necessary.
  Interventions: Device: ExAblate MR-guided Focused Ultrasound Bilateral Anterior Capsulotomy
- Sham FUS (Sham Comparator): The sham procedure will be identical in planning and execution to the ExAblate procedure with the only exception being that the energy output will be 0 for the sham-treated subjects. To perform the sham treatment, the sonication will be performed with energy output disabled. For sham subjects, the physician will interact with a subject in a similar manner and for a similar duration to simulate an actual procedure. When possible, the treating physician may determine a sonication (treatment) time for sham subjects to be similar to that which is occurring in the ExAblate procedure to maintain consistency between treatment arms. It should be noted that all treatment times of both treatment arms will be captured in the study CRF.
  Interventions: Device: ExAblate MR-guided Focused Ultrasound Bilateral Anterior Capsulotomy

INTERVENTIONS:
Device: ExAblate MR-guided Focused Ultrasound Bilateral Anterior Capsulotomy — The ExAblate transcranial system combines a focused ultrasound surgery delivery system and a conventional diagnostic 3T MRI scanner. The ExAblate transcranial system provides real-time therapy planning algorithm, thermal dosimetry, and closed-loop therapy control.

SUMMARY:
The goal of this clinical trial is to determine if ExAblate MR-guided Focused Ultrasound (MRgFUS) bilateral anterior capsulotomy can be used safely and effectively to relieve symptoms of moderate to severe obsessive compulsive disorder (OCD) in individuals who have not benefited from psychotherapy and medications.

The main questions it aims to answer are:

1. Can ExAblate MRgFUS capsulotomy be safely delivered to individuals suffering from treatment-refractory OCD through an intact skull with a risk and side-effect profile that is comparable to other neurosurgical approaches for capsulotomy?
2. Will ExAblate MRgFUS capsulotomy result in improvement in clinical symptoms and quality of life metrics that are similar to those seen with other surgical approaches for capsulotomy?

In the first stage of the study, participants with severe, treatment resistant OCD (n=10) will be recruited in two centers (Harvard and Stanford) and treated with best medical care (BMT) for 6 months. Thereafter, they will receive the ExAblate MRgFUS procedure and then another BMT for 12 months. In the second stage of the study, participants with moderate to severe OCD (n=56) will be recruited in a multi-center study and treated with BMT plus real or sham MRgFUS for 12 months. Thereafter, those who received sham MRgFUS and did not improve will receive real MRgFUS and then treated with BMT for another 12 months.

DETAILED DESCRIPTION:
The proposed study aims to establish the safety and efficacy of ExAblate MR-guided Focused Ultrasound (MRgFUS) for patients with treatment-refractory obsessive-compulsive disorder (OCD). Bilateral anterior thermo-capsulotomy and gamma-knife capsulotomy are well-known and effective treatments for treatment-refractory OCD patients. In this study, the investigators will use the ExAblate MRgFUS technology (Insightec Ltd) as a new method for capsulotomy for OCD patients. The ExAblate MRgFUS technology for neuro-related clinical applications has received FDA approval for Essential Tremor. In addition, the FDA approved an expansion of the ExAblate Neuro to include the treatment of tremor-dominant Parkinson's Disease. The study is designed to demonstrate safety and effectiveness and intended as a primary clinical support for a future marketing application.

The investigators propose a two-stage research protocol to establish the safety and efficacy of ExAblate MRgFUS for patients with treatment-resistant OCD. The first stage will be designed as a 'patient as own control' paradigm. Severe, treatment resistant OCD patients (n=10) will be recruited in two centers (Harvard and Stanford) and treated for 6 months by a best medical treatment (BMT) protocol followed by the ExAblate MRgFUS procedure plus BMT for another 12 months. The second stage will be designed as a 'double blind randomized control trial' paradigm. Moderate to severe, partially treatment resistant OCD patients (n=56) will be recruited in a multi-centered study and randomized into the ExAblate MRgFUS or sham procedures. They will be treated by BMT plus MRgFUS or BMT plus sham for 12 months followed by BMT plus the Exablate MRgFUS for the non-responding sham group for another 12 months.

This study is the first to evaluate ExAblate MRgFUS for OCD in the USA. This protocol was developed by two collaborating centers at Harvard and Stanford Universities, with two experienced and dedicated multidisciplinary teams of psychiatrists, neurosurgeons, psychologists, radiologists and neurologists. The suggested technical protocol using the ExAblate MRgFUS system for OCD is derived from a reported Korean study and an on-going Canadian clinical study.

The study is funded by the Focused Ultrasound Foundation and Insightec Ltd.

ELIGIBILITY:
Inclusion Criteria:

1. 25-64 years, inclusive.
2. Patients who are able and willing to give consent and able to attend study visits, as determined by both study psychiatrist and the surgeon.
3. DSM-5 diagnosis of Obsessive-Compulsive Disorder (OCD), at least 5-year illness history, with a minimum score of 28 on the Yale-Brown Obsessive Compulsive Scale (Y-BOCS) for stage I and a minimum score of 24 on Y-BOCS for stage II.
4. Medication-refractoriness as determined by an adequate dose and duration of standard psychiatric treatments (including psychotherapy and/or pharmacology) as determined by psychiatrists associated with the study. Including specifically:

   1. Failed adequate trial of three or more medications accepted as first line in the treatment of OCD such as selective serotonin reuptake inhibitors (SSRIs, e.g. fluoxetine, citalopram), selective serotonin-norepinephrine reuptake inhibitors (SNRIs), tricyclic antidepressants (TCAs, e.g. clomipramine) or other antidepressants at the maximal tolerated dose. Adequate maximal doses and minimal duration of these medication are listed in Table 2 below.
   2. Attempted augmentation, if tolerated, by at least two medications known to be second line treatments for OCD such as clonazepam, haloperidol, risperidone, olanzapine, gabapentin.
   3. An adequate trial of cognitive behavioral therapy (CBT) delivered by a therapist experienced in treating OCD. Criteria for an adequate CBT are listed in Table 3 below.
   4. In stage II patients that cannot tolerate pharmacotherapy or participate in psychotherapy will be included in the study.
5. A consistent dose of all medications in the 30 days prior to study entry
6. Able to communicate sensations during the ExAblate MRgFUS treatment

Exclusion Criteria:

1. Presence of significant cognitive impairment (as measured by a score <25 on the mini-mental state examination, MMSE)
2. Lifetime diagnosis of psychosis or bipolar disorder or presence of suicidality (as measured by a score >=2, item 9 of the BDI or high suicidal risk measured by the Columbia Suicide Severity Rating Scale (C-SSRS)). Subjects with stable, chronic anxiety or depressive disorders may be included provided their medications have been stable for at least 3 months prior to study entry and if deemed appropriately managed by the site psychiatrist.
3. DSM-5 diagnosis of substance use disorder (SUD) within the past 6 months
4. Patients with unstable cardiac status [e.g. unstable angina pectoris on medication; patients' medication (other than diuretic); patients on anti-arrhythmic drugs; severe hypertension (diastolic BP > 100 on medication)]
5. Cerebrovascular disease (e.g. CVA within 6 months), history of intracranial hemorrhage or intracranial aneurysms requiring treatment or arterial venous malformations (AVMs) requiring treatment
6. Untreated, uncontrolled sleep apnea
7. Patients with brain tumors, epilepsy, neurodegenerative disease or any other major neurological disorder
8. Patients with standard contraindications for MR imaging such as non-MRI compatible implanted metallic devices including cardiac pacemakers, size limitations, etc.
9. Known intolerance or allergies to MRI contrast agent (e.g. Gadolinium or Magnevist) including advanced kidney disease
10. Subjects who weigh more than the upper weight limit of the MR scanner table and who cannot fit into the MR scanner
11. An Overall Skull Density Ratio of less than 0.40 as calculated from the screening CT
12. Severely impaired renal function (estimated glomerular filtration rate < 30ml/min/1.73 m2) or receiving dialysis
13. Laboratory biochemical evidence of abnormal bleeding and/or coagulopathy, including risk factors for intraoperative or postoperative bleeding (platelet count less than 100,000 per cubic millimeter or abnormal INR)
14. Current medical condition resulting in abnormal bleeding and/or coagulopathy.
15. Receiving anticoagulant (e.g. warfarin) or antiplatelet (e.g. aspirin) therapy within one week of focused ultrasound procedure or drugs known to increase risk of hemorrhage (e.g. Avastin) within one month of focused ultrasound procedure. Receiving medications or supplements that increase the risk of bleeding such as NSAIDS, Ginko Baloba and Ginseng within one week of focused ultrasound procedure.
16. Individuals who are not able or willing to tolerate the required prolonged stationary supine position during treatment
17. Are participating or have participated in another clinical trial in the last 30 days
18. Patients unable to communicate with the investigator and staff
19. Currently pregnant (as determined by history and serum HCG) or lactating
20. Life-threatening systemic disease that include and not limited to the following will be excluded from the study participation: HIV, liver failure, blood dyscrasias, etc.

Ages: 25 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 66 (Estimated)
Dates: Start 2026-04 (Estimated); Primary Completion 2030-06 (Estimated); Study Completion 2032-06 (Estimated)

PRIMARY OUTCOMES:
Yale-Brown Obsessive-Compulsive Scale (YBOCS) | 12 months
  clinical scale specific to obsessive-compulsive disorder

SECONDARY OUTCOMES:
Clinical Global Impression (CGI) scale | 12 months
World Health Organization Disability Assessment Schedule 2.0 (WHODAS 2.0) | 12 months
  disability measure
Hamilton Rating Scale for Depression (HAM-D) | 12 months
  Clinician-rated depression scale
Hamilton Rating Scale for Anxiety (HAM-A) | 12 months
  Clinician-rated anxiety scale
Beck Depression Inventory (BDI) | 12 months
  Self-administered depression rating scale
Beck Anxiety Inventory (BAI) | 12 months
  Self-administered anxiety rating scale
Evaluation of the incidence and severity of procedure related complications | 12 months
  Subjective assessment of safety
Quality-of-Life Enjoyment and Satisfaction Questionnaire (QLESQ) | 12 months
  quality of life assessment

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Stanford University, Palo Alto, California
  - Brigham and Women's Hospital, Boston, Massachusetts

IPD SHARING:
Plan to Share IPD: Undecided